CLINICAL TRIAL: NCT02208947
Title: Consumer Engagement to Increase Advance Care Planning
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: failure to accure
Sponsor: University of Pittsburgh (Other)
Collaborators: Donaghue Medical Research Foundation (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Amber Barnato, MD, MPH, MS, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRO13120230
Record Dates: First submitted 2014-06-19; First posted 2014-08-05 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Advance Care Planning
Keywords: advance care planning; decision making; patient engagement; patient education; financial incentives; behavioral economics
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PREPARE (Active Comparator): Partnership HealthPlan of California (PHC) pays primary care physicians (PCPs) to discuss and document ACP with Medi-Cal beneficiaries aged 65 and older and those younger than 65 with a life-limiting illness (usual care). The control condition, or "enhanced usual care," adds a packet of educational information about ACP and access to the PREPARE website and verbal encouragement by their PCP delivered during a routine clinic visit to usual care.
  Interventions: Behavioral: PREPARE
- PREPARE + consumer financial incentive (Experimental): The experimental condition adds a consumer-directed financial incentive to enhanced usual care (provider-directed financial incentive and educational packet with information about the PREPARE website). Specifically, subjects will receive an immediate financial reward upon completing self-directed ACP (e.g., PREPARE steps 1-4) and a small probability of a large reward for discussing the plans with their physician (e.g., PREPARE step 5, documented by the PHC ACP attestation form).
  Interventions: Behavioral: Consumer financial incentive; Behavioral: PREPARE

INTERVENTIONS:
Behavioral: Consumer financial incentive — Immediate financial reward upon completing self-directed ACP (e.g., completing the web-based educational modules on PREPARE steps 1-4) and a small probability of a large reward for discussing the plans with their physician (e.g., PREPARE step 5, documented by the PHC ACP attestation form).
  Arms: PREPARE + consumer financial incentive
Behavioral: PREPARE — PREPARE for your care is 5-step on-line ACP process developed specifically for low-literacy Medi-Cal populations. PREPARE can be navigated as interactive, self-directed modules or "played" like a movie, at a time or a place of the subject's own choosing (e.g., home, work, public library).

SUMMARY:
The specific aims of the project are: 1) to test the effectiveness of consumer-directed financial incentives paired with provider-directed financial incentives, compared to provider-directed financial incentives alone, for increasing advance care planning (ACP) among Medicaid beneficiaries; and 2) to assess perceptions regarding the appropriateness of consumer-directed financial incentives for ACP among study participants. The investigators hypothesize that consumer-directed financial incentives will result in a 15-percentage point absolute increase in the proportion of subjects completing ACP. The investigators do not advance hypotheses about the qualitative component.

DETAILED DESCRIPTION:
This is a parallel cluster randomized controlled single-blind trial of consumer-directed financial incentives paired with provider-directed financial incentives (intervention), compared to provider-directed financial incentives alone (control) on the completion of ACP among Partnership HealthPlan of California (PHC) Medi-Cal patients. PHC is a county-organized health system contracted by the State of California to provide a health care delivery system for 360,000 Medi-Cal beneficiaries in Northern California. PHC has 400 contracted Primary Care Provider (PCP) entities, representing over 2000 individual physicians, working in solo practice, small groups, community health centers, large groups, and integrated health systems. The rationale for using PHC is their commitment to experimenting with strategies to improve ACP, including their current quality improvement program incentive payment to PCPs to discuss and document ACP with patients 65+ and <65 with a serious chronic illness.

The investigators will randomize 40 PCPs to one of two different patient education packets for their patients. Each PCP is eligible for financial incentives for documenting ACP (usual care), regardless of the randomization group.

Each PCP will be responsible for identifying and enrolling 10 eligible subjects during routine clinic visits, for a target enrollment of 400 patient subjects.

The investigators will stratify randomization based on salience of the financial incentive (e.g., accrues directly to non-salaried provider, such as in a private practice, or accrues to the organization of a salaried provider, such as in a Federally Qualified Health Center or multispecialty group).

All enrolled patients will receive access to the patient education tool, Prepare for Your Care (www.prepareforyourcare.org), developed by Dr. Sudore for low-literacy Medi-Cal populations, in their education packets. The intervention group patients will additionally be offered a consumer (patient) financial incentive. the primary outcome of the study is having a conversation with the PCP about ACP. Secondary outcomes include: 1) website use metrics and 2) attitudes about providing financial incentives for ACP (among a purposively sampled subset of participants).

ELIGIBILITY:
PCP Subject Inclusion Criteria:

* Partnership HealthPlan of California Medicaid and/or Medicare provider

PCP Subject Exclusion Criteria:

* Prohibition by clinic director

Patient Subject Inclusion Criteria:

* Partnership HealthPlan of California Medicaid and/or Medicare enrollee;
* Age 65+ or < 65 with a life-limiting illness (including advanced cardiac disease [end-stage congestive heart failure, severe coronary artery disease, cardiomyopathy (LVEF <25%)], advanced chronic obstructive pulmonary disease, amputation due to vascular disease, cancer [metastatic/recurrent], dementia, diabetes mellitus with creatinine clearance under 50, or an amputation, end stage renal disease, generalized debility and decreased functioning, long term resident of skilled nursing facility, stroke [w/at least 50% decreased function]);
* Internet access (computer, tablet, phone)

Patient Subject Exclusion Criteria:

* Completion of a Partnership HelathPlan of California advance care planning attestation form within the last 12 months;
* Inability to read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Advance care planning conversation with provider | 2 months (+/- 1 month)
  The primary outcome is the patient discussing their ACP with their provider within 2 months of having received the study advance care planning information packet, measured by the provider submitting an attestation form to Partnership HealthPlan of California to receive their ACP quality incentive payment.

SECONDARY OUTCOMES:
Use of the PREPARE website | 2 months (+/- 1 month)
  The process measure is developing a plan using the PREPARE website, measured by tracking website user metrics and receipt of the subject's "action plan and summary" by e-mail.

CONTACTS AND LOCATIONS:
Overall Officials: Amber E Barnato, MD MPH MS, Principal Investigator — University of Pittsburgh
Locations (1):
- Partnership HealthPlan-contracting provider groups in Northern California, Fairfield, California, United States